CLINICAL TRIAL: NCT01125189
Title: A Phase 2b Study of Daclatasvir in Combination With Peg-Interferon Alfa-2a and Ribavirin in Treatment Naive Subjects With Chronic Hepatitis C Genotype 1 and 4 Infection
Brief Title: Study of Daclatasvir (BMS-790052) Add-on to Standard of Care in Treatment- naïve Patients
Acronym: HEPCAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI444-010; 2010-018295-24 (EudraCT Number)
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Results first posted 2015-10-23 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Daclatasvir plus peg-interferon alfa-2a and ribavirin (20 mg) (Experimental)
  Interventions: Drug: Daclatasvir; Drug: peg-interferon alfa-2a; Drug: ribavirin
- Daclatasvir plus peg-interferon alfa-2a and ribavirin (60 mg) (Experimental)
  Interventions: Drug: Daclatasvir; Drug: peg-interferon alfa-2a; Drug: ribavirin
- Placebo plus peg-interferon alfa-2a and ribavirin (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: peg-interferon alfa-2a; Drug: ribavirin

INTERVENTIONS:
Drug: Daclatasvir — Tablets, oral, 20 mg, once daily, 12-24 weeks, depending on response
  Arms: Daclatasvir plus peg-interferon alfa-2a and ribavirin (20 mg)
Drug: Daclatasvir — Tablets, oral, 60 mg, once daily, 12-24 weeks, depending on response
  Arms: Daclatasvir plus peg-interferon alfa-2a and ribavirin (60 mg)
Drug: Placebo — Tablets, oral, 0 mg, once daily, 24 weeks
  Arms: Placebo plus peg-interferon alfa-2a and ribavirin
Drug: peg-interferon alfa-2a — Syringe, subcutaneous Injection, 180 µg, once weekly, 24 or 48 weeks depending on response
  Other Names: Pegasys
Drug: ribavirin — Tablets, oral, 1000 or 1200 mg based on weight, once daily, 24 or 48 weeks depending on response
  Other Names: Copegus

SUMMARY:
To establish that at least 1 dose of daclatasvir combined with standard of care (pegylated interferon and ribavirin) is safe and well tolerated and demonstrates extended rapid virologic response rates at least 35% greater than those with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients chronically infected with hepatitis C virus (HCV) genotype 1 or 4
* HCV RNA viral load of ≥100,000 IU/mL
* No previous exposure to interferon, pegIFNα, or RBV
* Results of a liver biopsy demonstrating absence of cirrhosis obtained ≤24 months prior to randomization. Compensated cirrhotics with Hepatitis C virus genotype 1 infection are eligible, but will be capped at 10% of the randomized study population (biopsy can be from any time period prior to randomization)
* Findings on ultrasound, computed tomography scan, or magnetic resonance imaging 12 months prior to randomization that do not demonstrate evidence of hepatocellular carcinoma
* Body mass index of 18 to 35 kg/m^2

Exclusion Criteria:

* Positive for hepatitis B or HIV-1/HIV-2 antibody at screening
* Evidence of a medical condition associated with chronic liver disease other than HCV
* Evidence of decompensated cirrhosis based on radiologic criteria or biopsy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2010-07; Primary Completion 2012-04 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (64):
- United States (33):
  - Alabama Liver & Digestive Specialists (Alds), Montgomery, Alabama
  - Scripps Clinic, La Jolla, California
  - Cli, Los Angeles, California
  - Desta Digestive Disease Medical Center, San Diego, California
  - University Of California, San Francisco/Sf General Hospital, San Francisco, California
  - California Pacific Medical Center, San Francisco, California
  - Kaiser Permanente Medical Center, San Francisco, California
  - Transplant Center And Hepatology Clinic, B-154, Aurora, Colorado
  - Yale University School Of Medicine, New Haven, Connecticut
  - University Of Florida Hepatology, Gainesville, Florida
  - University Of Miami, Miami, Florida
  - Miami Research Associates, South Miami, Florida
  - Indiana University, Indianapolis, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Digestive Disease Associates, P.A., Baltimore, Maryland
  - Johns Hopkins University, Lutherville, Maryland
  - Claudia T. Martorell, Md, Llc, Springfield, Massachusetts
  - James Sungsik Park, M.D. C.N.S.C., Great Neck, New York
  - Upper Delaware Valley Infectious Diseases, Pc, Monticello, New York
  - James J Peters Vamc, The Bronx, New York
  - University Of North Carolina At Chapel Hill School Of Med, Chapel Hill, North Carolina
  - Carolinas Center For Liver Disease, Statesville, North Carolina
  - Options Health Research, Llc, Tulsa, Oklahoma
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - University Of Pennsylvania, Philadelphia, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Nashville Medical Research Institute, Nashville, Tennessee
  - North Texas Research Institute, Arlington, Texas
  - St. Luke'S Episcopal Hospital - Baylor College Of Medicine, Houston, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Metropolitan Research, Fairfax, Virginia
  - Dean Clinic, Madison, Wisconsin
- Australia (6):
  - Local Institution, Darlinghurst, New South Wales
  - Local Institution, Westmead Nsw, New South Wales
  - Local Institution, Woolloongabba, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Clayton Vic, Victoria
  - Local Institution, Camperdown
- Canada (5):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Victoria, British Columbia
  - Local institution, Toronto, Ontario
  - Local Institution, Toronto, Ontario
- Denmark (3):
  - Local Institution, Aarhus
  - Local Institution, Hvidovre
  - Local Institution, Odense
- Egypt (2):
  - Local Institution, Shebin Elkom, Monufia Governorate
  - Local Institution, Cairo
- France (5):
  - Local Institution, Créteil
  - Local Institution, Marseille
  - Local Institution, Montpellier
  - Local Instituition, Paris
  - Local Institution, Paris
- Germany (4):
  - Local Institution, Düsseldorf
  - Local Institution, Essen
  - Local Institution, Frankfurt
  - Local Institution, Hamburg
- Italy (2):
  - Local Institution, Cisanello (pisa)
  - Local Institution, Pavia
- Local Institution, Guadalajara, Jalisco, Mexico
- Local Institution, San Juan, Puerto Rico
- Sweden (2):
  - Local Institution, Gothenburg
  - Local Institution, Stockholm

REFERENCES:
- [Derived] Hezode C, Hirschfield GM, Ghesquiere W, Sievert W, Rodriguez-Torres M, Shafran SD, Thuluvath PJ, Tatum HA, Waked I, Esmat G, Lawitz EJ, Rustgi VK, Pol S, Weis N, Pockros PJ, Bourliere M, Serfaty L, Vierling JM, Fried MW, Weiland O, Brunetto MR, Everson GT, Zeuzem S, Kwo PY, Sulkowski M, Brau N, Hernandez D, McPhee F, Wind-Rotolo M, Liu Z, Noviello S, Hughes EA, Yin PD, Schnittman S. Daclatasvir plus peginterferon alfa and ribavirin for treatment-naive chronic hepatitis C genotype 1 or 4 infection: a randomised study. Gut. 2015 Jun;64(6):948-56. doi: 10.1136/gutjnl-2014-307498. Epub 2014 Jul 30. PMID 25080450
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 64 sites in 11 countries.
Pre-assignment Details: A total of 558 participants were enrolled in this study, and 395 participants were randomized and treated.
Groups:
- Daclatasvir (20 mg) + Peg-interferon Alfa-2a + Ribavirin: Participants received daclatasvir tablets 20 mg orally, once daily with pegylated-interferon alfa-2a solution for injection 180 µg per 0.5 mL subcutaneously, once weekly, and ribavirin tablets 1000-1200 mg orally, twice daily for a total duration of 12 weeks. After Week 12, additional treatment was provided with interferon and ribavirin for a total of 24 or 48 weeks of therapy depending on whether or not the participant achieved an on-treatment response as defined in protocol.
- Daclatasvir (60 mg) + Peg-interferon Alfa-2a + Ribavirin: Participants received daclatasvir tablets 60 mg orally, once daily with pegylated-interferon alfa-2a solution for injection 180 µg per 0.5 mL subcutaneously, once weekly, and ribavirin tablets 1000-1200 mg orally, twice daily for a total duration of 12 weeks. After Week 12, additional treatment was provided with interferon and ribavirin for a total of 24 or 48 weeks of therapy depending on whether or not the participant achieved an on-treatment response as defined in protocol.
- Placebo + Peg-interferon Alfa-2a + Ribavirin: Participants received placebo matched with daclatasvir tablets orally, once daily with pegylated-interferon alfa-2a solution for injection 180 µg per 0.5 mL subcutaneously, once weekly, and ribavirin tablets 1000-1200 mg orally, twice daily, for a total duration of 24 weeks and pegylated-interferon alfa-2a and ribavirin, for a total duration of 48 weeks.
Period: Treatment Period
Arm/Group | Daclatasvir (20 mg) + Peg-interferon Alfa-2a + Ribavirin | Daclatasvir (60 mg) + Peg-interferon Alfa-2a + Ribavirin | Placebo + Peg-interferon Alfa-2a + Ribavirin
Started | 159 | 158 | 78
Completed | 128 | 123 | 37
Not Completed | 31 | 35 | 41
Not completed — Lack of Efficacy | 15 | 18 | 25
Not completed — Adverse Event | 7 | 8 | 8
Not completed — Withdrawal by Subject | 3 | 1 | 1
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Poor compliance/noncompliance | 0 | 1 | 0
Not completed — Participants requested to discontinue | 1 | 3 | 4
Not completed — Other reasons | 1 | 1 | 0
Not completed — Completed 24 week treatment period only | 2 | 1 | 2
Period: Follow up Period
Arm/Group | Daclatasvir (20 mg) + Peg-interferon Alfa-2a + Ribavirin | Daclatasvir (60 mg) + Peg-interferon Alfa-2a + Ribavirin | Placebo + Peg-interferon Alfa-2a + Ribavirin
Started | 152 (All participants who received treatment continued in the follow-up phase.) | 153 (All participants who received treatment continued in the follow-up phase.) | 74 (All participants who received treatment continued in the follow-up phase.)
Completed | 132 | 138 | 58
Not Completed | 20 | 15 | 16
Not completed — Withdrawal by Subject | 3 | 2 | 5
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 12 | 9 | 6
Not completed — Other reasons | 4 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daclatasvir (20 mg) + Peg-interferon Alfa-2a + Ribavirin | Daclatasvir (60 mg) + Peg-interferon Alfa-2a + Ribavirin | Placebo + Peg-interferon Alfa-2a + Ribavirin | Total
Number analyzed (Participants) | 159 | 158 | 78 | 395
Age, Customized [Number; unit: participants]
  <65 years | 154 | 154 | 77 | 385
  ≥65 years | 5 | 4 | 1 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 55 | 23 | 130
  Male | 107 | 103 | 55 | 265
Hepatitis C Virus RNA Distribution [Number; unit: participants]
  <800,000 IU/mL | 26 | 35 | 17 | 78
  ≥800,000 IU/mL | 133 | 123 | 61 | 317
IL-28B Genotype [Number; unit: participants]
  CC genotype | 53 | 44 | 23 | 120
  CT genotype | 82 | 86 | 38 | 206
  TT genotype | 17 | 18 | 11 | 46
  Missing | 7 | 10 | 6 | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Hepatitis C Virus (HCV) Genotype 1 Participants With Extended Rapid Virologic Response (eRVR)
Description: eRVR was defined as HCV RNA <lower limit of quantitation and target not detected at both Weeks 4 and 12 on treatment.
Time Frame: Weeks 4 and 12
Population: All treated participants. Here, 'number of participants' analyzed (N) signifies number of participants evaluable for this outcome measure.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Daclatasvir (20 mg) + Peg-interferon Alfa-2a + Ribavirin | Daclatasvir (60 mg) + Peg-interferon Alfa-2a + Ribavirin | Placebo + Peg-interferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 147 | 146 | 72
percentage of participants | 54.4 [49.2 to 59.7] | 54.1 [48.8 to 59.4] | 13.9 [8.7 to 19.1]

2. Primary Outcome: Percentage of Hepatitis C Virus (HCV) Genotype 1 Participants With Sustained Virologic Response (SVR24)
Description: SVR24 was defined as HCV <lower limit of quantitation (LLOQ) and target not detected (TND) at follow-up Week 24. The LLOQ was 25 IU/mL, and <LLOQ, TND was 10 IU/mL. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory.
Time Frame: Follow-up Week 24
Population: All treated participants. Here, N signifies number of participants evaluable for this outcome measure.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Daclatasvir (20 mg) + Peg-interferon Alfa-2a + Ribavirin | Daclatasvir (60 mg) + Peg-interferon Alfa-2a + Ribavirin | Placebo + Peg-interferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 147 | 146 | 72
percentage of participants | 59.2 [54.0 to 64.4] | 59.6 [54.4 to 64.8] | 37.5 [30.2 to 44.8]

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs), Discontinuations Due to Adverse Events (AEs), and Who Died
Description: SAE was defined as a medical event that at any dose resulted in death, persistent or significant disability/incapacity, or drug dependency/abuse; was life threatening, an important medical event, or a congenital anomaly/birth defect; or required or prolonged hospitalization.
Time Frame: From start of study treatment (day 1) up to follow-up Week 48
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Daclatasvir (20 mg) + Peg-interferon Alfa-2a + Ribavirin | Daclatasvir (60 mg) + Peg-interferon Alfa-2a + Ribavirin | Placebo + Peg-interferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 159 | 158 | 78
participants
  SAEs | 12 | 13 | 6
  Discontinuations Due to AEs | 7 | 7 | 8
  Death | 2 | 0 | 0

4. Secondary Outcome: Percentage of Hepatitis C Virus (HCV) Genotype 1 Participants With Rapid Virologic Response (RVR)
Description: RVR was defined as undetectable RNA (HCV RNA <lower limit of quantitation [LLOQ], target not detected [TND]) at Week 4. The LLOQ was 25 IU/mL, and <LLOQ, TND was 10 IU/mL. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory. N=Number of participants analyzed for this outcome.
Time Frame: Week 4
Population: All treated participants. Here, N signifies number of participants evaluable for this outcome measure.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Groups:
- Daclatasvir (20 mg) + Peg-interferon Alfa-2a + Ribavirin: Participants received daclatasvir tablets 20 mg orally, once daily with pegylated--interferon alfa-2a solution for injection 180 µg per 0.5 mL subcutaneously, once weekly, and ribavirin tablets 1000-1200 mg orally, twice daily for a total duration of 12 weeks. After Week 12, additional treatment was provided with interferon and ribavirin for a total of 24 or 48 weeks of therapy depending on whether or not the participant achieved an on-treatment response as defined in protocol.
Arm/Group | Daclatasvir (20 mg) + Peg-interferon Alfa-2a + Ribavirin | Daclatasvir (60 mg) + Peg-interferon Alfa-2a + Ribavirin | Placebo + Peg-interferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 147 | 146 | 72
percentage of participants | 59.9 [54.7 to 65.0] | 56.8 [51.6 to 62.1] | 15.3 [9.8 to 20.7]

5. Secondary Outcome: Percentage of Hepatitis C Virus (HCV) Genotype 1 Participants With Complete Early Virologic Response (cEVR)
Description: cEVR was defined as undetectable RNA (HCV RNA <lower limit of quantitation [LLOQ], target not detected [TND]) at Week 12. The LLOQ was 25 IU/mL, and <LLOQ, TND was 10 IU/mL. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory. N=Number of participants analyzed for this outcome.
Time Frame: Week 12
Population: All treated participants. Here, N signifies number of participants evaluable for this outcome measure.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Groups:
- Placebo + Peg-interferon Alfa-2a + Ribavirin: Participants received placebo matched with daclatasvir tablets orally, once daily with pegylate--interferon alfa-2a solution for injection 180 µg per 0.5 mL subcutaneously, once weekly, and ribavirin tablets 1000-1200 mg orally, twice daily, for a total duration of 24 weeks and pegylated-interferon alfa-2a and ribavirin, for a total duration of 48 weeks.
Arm/Group | Daclatasvir (20 mg) + Peg-interferon Alfa-2a + Ribavirin | Daclatasvir (60 mg) + Peg-interferon Alfa-2a + Ribavirin | Placebo + Peg-interferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 147 | 146 | 72
percentage of participants | 77.6 [73.1 to 82.0] | 75.3 [70.8 to 79.9] | 43.1 [35.6 to 50.5]

6. Secondary Outcome: Percentage of Hepatitis C Virus (HCV) Genotype 1 Participants With 12-week Sustained Virologic Response (SVR12)
Description: SVR12 was defined as undetectable RNA (HCV RNA < lower limit of quantitation (LLOQ), target not detected (TND) at follow-up Week 12. The LLOQ was 25 IU/mL, and <LLOQ, TND was 10 IU/mL. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory. N=Number of participants analyzed for this outcome.
Time Frame: Follow-up Week 12
Population: All treated participants. Here, N signifies number of participants evaluable for this outcome measure.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Groups:
- Daclatasvir (60 mg) + Peg-interferon Alfa-2a + Ribavirin: Participants received daclatasvir tablets 60 mg orally, once daily with pegylated--interferon alfa-2a solution for injection 180 µg per 0.5 mL subcutaneously, once weekly, and ribavirin tablets 1000-1200 mg orally, twice daily for a total duration of 12 weeks. After Week 12, additional treatment was provided with interferon and ribavirin for a total of 24 or 48 weeks of therapy depending on whether or not the participant achieved an on-treatment response as defined in protocol.
Arm/Group | Daclatasvir (20 mg) + Peg-interferon Alfa-2a + Ribavirin | Daclatasvir (60 mg) + Peg-interferon Alfa-2a + Ribavirin | Placebo + Peg-interferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 147 | 146 | 72
percentage of participants | 64.6 [59.6 to 69.7] | 60.3 [55.1 to 65.5] | 36.1 [28.9 to 43.4]

7. Secondary Outcome: Percentage of Resistant Variants Associated With Virologic Failure
Description: Virologic failure was defined as:
  1. Virologic breakthrough: confirmed >1 log10 increase in hepatitis C virus (HCV) RNA over nadir or confirmed RNA ≥lower limit of quantitation (LLOQ) after confirmed HCV RNA <LLOQ, target not detected (TND) while on treatment
  2. <1 log10 decrease in HCV RNA from baseline at Week 4 of treatment
  3. Failure to achieve early virologic response: <2 log10 decrease in HCV RNA from baseline and HCV RNA ≥LLOQ at Week 12 of treatment
  4. HCV RNA < LLOQ, TD or ≥ LLOQ at Week 12 and ≥ LLOQ at Week 24
  5. HCV RNA ≥LLOQ or <LLOQ, target detected (TD) at the end of treatment (EOT) (including early discontinuation)
  6. Relapse, defined as HCV RNA ≥LLOQ or <LLOQ, TD during follow-up, after HCV RNA < LLOQ, TND at EOT.
  The LLOQ was 25 IU/mL, and <LLOQ, TND was 10 IU/mL. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory. N=Number of participants analyzed for this outcome.
Time Frame: Follow-up Week 48
Population: All treated participants. Here, N signifies number of participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Daclatasvir (20 mg) + Peg-interferon Alfa-2a + Ribavirin | Daclatasvir (60 mg) + Peg-interferon Alfa-2a + Ribavirin | Placebo + Peg-interferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 147 | 146 | 72
percentage of participants
  Virologic Breakthrough | 8.2 | 10.3 | 2.8
  Week 4 Futility Rule | 2.0 | 2.1 | 25.0
  Detectable HCV RNA at EOT | 7.5 | 6.8 | 5.6
  Other Criteria | 1.4 | 0.1 | 6.9
  Relapse | 18.5 | 19.0 | 22.0

ADVERSE EVENTS:
Time Frame: From start of study treatment (day 1) up to 7 days post last dose of study treatment (Week 24)
Description: On-treatment period.
Groups:
- Daclatasvir (20 mg) + Peg-interferon Alfa-2a + Ribavirin: Participants received daclatasvir tablets 20 mg orally, once daily with pegylated--interferon alfa-2a solution for injection 180 µg per 0.5 mL subcutaneously, once weekly, and ribavirin tablets 1000-1200 mg orally, twice daily for a total duration of 12 weeks. After Week 12, additional treatment was provided with interferon and ribavirin for a total of 24 or 48 weeks of therapy depending on whether or not the patient achieved an on-treatment response as defined in protocol.
- Daclatasvir (60 mg) + Peg-interferon Alfa-2a + Ribavirin: Participants received daclatasvir tablets 60 mg orally, once daily with pegylated-interferon alfa-2a solution for injection 180 µg per 0.5 mL subcutaneously, once weekly, and ribavirin tablets 1000-1200 mg orally, twice daily for a total duration of 12 weeks. After Week 12, additional treatment was provided with interferon and ribavirin for a total of 24 or 48 weeks of therapy depending on whether or not the patient achieved an on-treatment response as defined in protocol.
Arm/Group | Daclatasvir (20 mg) + Peg-interferon Alfa-2a + Ribavirin | Daclatasvir (60 mg) + Peg-interferon Alfa-2a + Ribavirin | Placebo + Peg-interferon Alfa-2a + Ribavirin
Serious Adverse Events (participants affected / at risk) | 12/159 | 13/158 | 6/78
Other Adverse Events (participants affected / at risk) | 156/159 | 155/158 | 76/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daclatasvir (20 mg) + Peg-interferon Alfa-2a + Ribavirin (N=159) | Daclatasvir (60 mg) + Peg-interferon Alfa-2a + Ribavirin (N=158) | Placebo + Peg-interferon Alfa-2a + Ribavirin (N=78)
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Adjustment disorder (Psychiatric disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Death (General disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 1 | 0
Hypomania (Psychiatric disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Mental disorder (Psychiatric disorders) | 0 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1
Aplastic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Auricular perichondritis (Ear and labyrinth disorders) | 0 | 1 | 0
Carbuncle (Infections and infestations) | 0 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0
Electrocardiogram change (Investigations) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 1
Substance-induced psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Schizophrenia, paranoid type (Psychiatric disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daclatasvir (20 mg) + Peg-interferon Alfa-2a + Ribavirin (N=159) | Daclatasvir (60 mg) + Peg-interferon Alfa-2a + Ribavirin (N=158) | Placebo + Peg-interferon Alfa-2a + Ribavirin (N=78)
Anaemia (Blood and lymphatic system disorders) | 32 | 21 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 | 28 | 19
Asthenia (General disorders) | 18 | 14 | 7
Dry eye (Eye disorders) | 11 | 9 | 4
Dysgeusia (Nervous system disorders) | 13 | 12 | 4
Fatigue (General disorders) | 88 | 86 | 46
Injection site erythema (General disorders) | 10 | 12 | 5
Irritability (General disorders) | 35 | 37 | 22
Vision blurred (Eye disorders) | 7 | 6 | 7
Disturbance in attention (Nervous system disorders) | 5 | 7 | 6
Erythema (Skin and subcutaneous tissue disorders) | 9 | 5 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12 | 9 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 56 | 63 | 26
Sinusitis (Infections and infestations) | 11 | 3 | 3
Weight decreased (Investigations) | 12 | 8 | 8
Anxiety (Psychiatric disorders) | 15 | 15 | 6
Dry mouth (Gastrointestinal disorders) | 14 | 8 | 2
Memory impairment (Nervous system disorders) | 4 | 9 | 0
Nausea (Gastrointestinal disorders) | 56 | 53 | 20
Neutropenia (Blood and lymphatic system disorders) | 26 | 17 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 21 | 8
Constipation (Gastrointestinal disorders) | 8 | 11 | 3
Depression (Psychiatric disorders) | 24 | 21 | 10
Diarrhoea (Gastrointestinal disorders) | 36 | 37 | 14
Dry skin (Skin and subcutaneous tissue disorders) | 47 | 41 | 15
Dyspepsia (Gastrointestinal disorders) | 12 | 10 | 8
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 19 | 19 | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 11 | 2
Influenza like illness (General disorders) | 45 | 49 | 16
Insomnia (Psychiatric disorders) | 49 | 53 | 30
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 13 | 3
Decreased appetite (Metabolism and nutrition disorders) | 27 | 40 | 17
Dizziness (Nervous system disorders) | 22 | 24 | 9
Vomiting (Gastrointestinal disorders) | 19 | 15 | 11
Chest pain (General disorders) | 9 | 6 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 32 | 26 | 11
Headache (Nervous system disorders) | 68 | 68 | 36
Injection site rash (General disorders) | 2 | 4 | 6
Injection site reaction (General disorders) | 13 | 8 | 6
Rash (Skin and subcutaneous tissue disorders) | 54 | 40 | 25
Abdominal pain upper (Gastrointestinal disorders) | 8 | 9 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 39 | 41 | 13
Chills (General disorders) | 28 | 21 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 31 | 18
Myalgia (Musculoskeletal and connective tissue disorders) | 45 | 43 | 24
Abdominal pain (Gastrointestinal disorders) | 14 | 13 | 2
Depressed mood (Psychiatric disorders) | 3 | 10 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 7 | 4
Lower respiratory tract infection (Infections and infestations) | 2 | 1 | 4
Oral herpes (Infections and infestations) | 6 | 8 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 6 | 5
Pyrexia (General disorders) | 28 | 20 | 15
Sleep disorder (Psychiatric disorders) | 11 | 13 | 4
Upper respiratory tract infection (Infections and infestations) | 8 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.